CLINICAL TRIAL: NCT00553085
Title: Anxiety Disorders in Children - Association With Neurodevelopmental Delay/Disorder and Temperament/Personality. A Clinical Case-control Study
Brief Title: Anxiety Disorders in Children - Association With Neurodevelopmental Delay/Disorder
Status: Completed | Type: Observational
Sponsor: Regionsenter for barn og unges psykiske helse (Other)
Collaborators: The Research Council of Norway (Other); University Hospital, Akershus (Other); Lovisenberg Diakonale Hospital (Other); The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Hanne Kristensen, Director, Clinical Research Section, Regionsenter for barn og unges psykiske helse
Other Study IDs: 1.2006.2943; 181877/V50
Record Dates: First submitted 2007-11-02; First posted 2007-11-05 (Estimated); Last update posted 2014-06-20 (Estimated); Status verified 2014-06

CONDITIONS: Anxiety Disorders
Keywords: anxiety disorders; children; neurodevelopmental disorder; neurodevelopmental delay; temperament
MeSH Terms: conditions — Anxiety Disorders; Neurodevelopmental Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Saliva for measuring Cortisol
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Anx group
- ADHD group
- Nonanx/nonadhd group

SUMMARY:
The main objective of the study is to examine the relationship between anxiety disorders and neurodevelopmental disorder/delay in children aged 7- 13 years.

DETAILED DESCRIPTION:
Project summary Anxiety disorders (AD's) in childhood are common and may cause great suffering.Childhood AD's may persist into adulthood and knowledge of important risk factors for development and maintenance of these disorders is essential.The development of AD's is due to a complex interaction between biological and environmental factors.This study will examine the relationship between AD's and two biological risk factors:1.Neurodevelopmental delays/disorders (NDD'S) in motor and cognitive function and 2.Temperament/personality.To date a few studies have consistently found that motor impairment is associated with childhood anxiety and predicts persistent anxiety in adolescence.The association between AD's and NDD's in cognitive functions such as language and attention is far less studied. In contrast, there is a huge research literature on temperament as a risk factor for AD's.The temperamental trait "behavioural inhibition" has been shown to be particularly associated with AD's.However, very few studies have examined the interplay between NDD's, temperament and anxiety.The study is a clinical case-control study of children aged 7-13 years with AD's referred to three different out-patient clinics.The participants will be assessed by diagnostic interviews, neuropsychological tests and temperament/personality instruments.Comparison groups are:1.children with ADHD (to compare AD's with another mental disorder related to NDD's) and 2.Non-referred children without a mental disorder. Follow-up at 6 months,1 and 5 years.A pilot study at two of the three out-patient clinics to be included,showed a sufficient sample size.Anticipated implications of the study include increased knowledge of biological risk factors and of latent neurological brain correlates,as well as treatment implications.Children with NDD's are often met with demands they cannot cope with due to their neurodevelopmental immaturity.To adjust the demands to the child's actual level of functioning is important.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of anxiety disorder or ADHD or no diagnosis

Exclusion Criteria:

* Clinical diagnosis of PDD
* mental retardation
* children whose both parents do not speak Norwegian

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Consecutive patient sampling
Sampling Method: Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2007-09; Primary Completion 2009-12 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Diagnosis of anxiety disorder | 5 years

SECONDARY OUTCOMES:
Children's global assessment scale (CGAS) | 5 years
  The CGAS represents an assessment of the child's overall severity of disturbance with scores ranging from 1 (lowest functioning) to 100 (excellent functioning)

CONTACTS AND LOCATIONS:
Overall Officials: Hanne Kristensen, Ph.D., Principal Investigator — Regionsenter for barn og unges psykiske helse
Locations (2):
- Norway (2):
  - Akershus University Hospital, Lorenskog, Akershus
  - Lovisenberg Hospital, Oslo, Oslo County